CLINICAL TRIAL: NCT02745925
Title: Mechanism of Decreased Iron Absorption in Obesity: Controlling Adiposity-related Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: University of Monterrey, Mexico (Unknown)
Responsible Party: Principal Investigator, Isabelle Herter-Aeberli, Dr., Swiss Federal Institute of Technology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Fe_Abs_Ibu
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Obesity
Keywords: Iron bioavailability; Inflammation; Hepcidin; Iron absorption
MeSH Terms: conditions — Obesity; Inflammation | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- normal-weight (Experimental): normal-weight women
  Interventions: Drug: Ibuprofen
- obesity (Experimental): obese women
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen

SUMMARY:
The main iron regulatory protein in the human metabolism is hepcidin. In normal weight, healthy subjects, hepcidin is regulated through the iron status of the body: low iron status results in low hepcidin concentrations, which facilitates dietary iron absorption. In obesity, which is an inflammatory state, hepcidin concentrations are increased and iron absorption is reduced despite low iron stores, leading to iron deficiency over time. Whether lowering the chronic low-grade inflammation during a limited treatment period and thereby lowering hepcidin concentration can improve iron absorption is uncertain.

DETAILED DESCRIPTION:
In states of high hepcidin concentration, intestinal iron absorption (through enterocytes) and recycling of iron (through macrophages) is reduced. The extent to which non-heme iron is absorbed from the diet is influenced by the composition of the diet. Ascorbic acid is a potent enhancer of non-heme iron absorption. It's mechanism of action is luminal reduction of dietary ferric iron (Fe3+) to more soluble ferrous iron (Fe2+). A study in the inestigator's laboratory showed that the enhancing effect of ascorbic acid on non-heme iron absorption is reduced in overweight and obese individuals. Possible explanations for this fact are the different sites of action of ascorbic acid and serum hepcidin on the enterocytes in dietary iron absorption. Increased hepcidin reduces iron efflux into the circulation at the basolateral membrane of the enterocyte. Therefore the improved iron transport into enterocytes through ascorbic acid at the luminal side (via the divalent metal transporter (DMT)-1), by reducing Fe3+ to Fe2+ seems to be less successful. To improve iron absorption in obese subjects, an intervention at the basolateral membrane of the enterocyte would be needed.

ELIGIBILITY:
Inclusion Criteria:

* normal-weight (BMI18.5-24.9kg/m2) or obesity (BMI 29-40kg/m2)
* pre-menopausal
* no chronic illness and no significant medical conditions that could influence iron or inflammatory status other than obesity
* no-smoking

Exclusion Criteria:

* Diagnosed chronic disease or gastrointestinal disorders
* Metabolic disorders (e.g. diabetes)
* Regular use of medication (except oral contraceptives)
* Subject on a weight loss diet or planning to start a weight loss diet during the duration of the study
* Pregnancy or lactation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption | Days 15 and 45
  The fractional iron absorption from four test meals will be calculated based on the shift of the iron isotopic ratios in the collected blood samples 14 days after administration of the isotopically labeled meals. Calculation of fractional iron absorption will take into account the principles of isotope dilution and the fact that iron isotopic labels are not mono-isotopic. The investigators assumed iron incorporation into erythrocytes to be constant. Blood volume, needed for the calculation of fractional iron absorption will be estimated based on available data on blood volume estimations in obese women.

SECONDARY OUTCOMES:
Plasma ferritin | Days 1, 15, 30, 45
Hemoglobin | Days 1, 15, 30, 45
Transferrin receptor | Days 1, 15, 30, 45
Hepcidin | Days 1, 15, 30, 45
c-reactive protein | Days 1, 15, 30, 45
interleukin-6 | Days 1, 15, 30, 45
alpha-1-acid-glycoprotein | Days 1, 15, 30, 45

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Herter-Aeberli, PhD, Principal Investigator — University of Zurich
Locations (1):
- Human Nutrition Laboratory ETH Zurich, Zurich, Switzerland